CLINICAL TRIAL: NCT03274622
Title: Efficacy of Parent-implemented Treatment in Infant Siblings of Children With Autism Spectrum Disorder (ASD)
Brief Title: Efficacy of IMPACT in Infant Siblings of Children With ASD
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Paul Yoder, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 140924; 1R01DC013767-01 (NIH)
Record Dates: First submitted 2017-08-17; First posted 2017-09-07 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessors and coders are blind to treatment assignment. This will be achieved by using different people to conduct the treatment vs assessment and coding. Additionally, these different staff members have offices on different floors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impact Parent Training (Experimental): Parents receive 22 1.5-hour sessions with a Speech Language pathologist coaching them in the implementation of the Impact intervention
  Interventions: Behavioral: Impact Parent Training
- No Impact (Placebo Comparator): No parent coaching is provided
  Interventions: Behavioral: No Impact

INTERVENTIONS:
Behavioral: Impact Parent Training
  Arms: Impact Parent Training
Behavioral: No Impact
  Arms: No Impact

SUMMARY:
Over a 5 year period infant and baby siblings of children with autism spectrum disorders (ASD) will be recruited to this study and will be randomized into 2 groups. Parents of the intervention group will receive 12 weeks of coaching in how to implement this intervention. Parents randomized to the control group will not receive intervention coaching. Both groups will attend a series of clinic appointments for data collection that occur at 3 month intervals over a 9 month period.

DETAILED DESCRIPTION:
This two-site randomized controlled trail (RCT) will include a sample of 80 siblings of children with ASD (Sibs-ASD) (11 months, 15 days to 18 months, 15 days) who are stratified on initial cumulative-risk status for communication disorder and then randomly assigned to Ingersoll's Improving Parents As Communication Teachers (ImPACT; Ingersoll & Dvortcsak, 2010) treatment or to a business-as-usual (BAU) control condition. The following hypotheses will be tested:

1. Compared to the BAU Control, children assigned to the ImPACT group will show (a) more growth on pivotal skills and language level, and (b) a lesser degree of ASD symptomatology and language delay.
2. Pretreatment, cumulative-risk level will statistically interact with (i.e., moderate) treatment assignment to predict children's (a) change in pivotal skills and language, and (b) severity of autism symptoms and language delay.
3. Compared to the BAU Control, parents in ImPACT will have more optimal parenting stress and parenting efficacy, at least in parents with average or below average depressive symptoms prior to treatment (i.e., depressive symptoms will moderate the effect of ImPACT on parental stress and parenting efficacy).
4. The effect that ImPACT has on growth of pivotal skills and language will be mediated by parents' frequency and fidelity of use of ImPACT strategies at immediate post-treatment.
5. The effect of ImPACT on degree of children's language delay and ASD symptomatology at 6 months post-treatment will be mediated by their pivotal skill level at 3 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

Younger sibling of a child with ASD -

1. Age: 11 months, 15 days to 18 months, 15 days
2. Older biological sibling: Must have a diagnosis of Autism from UW or VU, which is confirmed via record review. If the older sibling was not diagnosed at UW or VU, then a diagnostic appointment must be made for the older sibling at the corresponding institution in order to confirm the diagnosis of ASD. Half-siblings are ok.
3. Vision - WNL corrected
4. Hearing - WNL corrected
5. Motor: The child must be able to sit independently while picking up objects and giving them to another person.

Exclusions:

No primary motor impairment. No feeding tubes. No other neurological or genetic conditions. Primary language exposure: The primary parent speak to the child using English 50% of the time, and process.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Growth in communication | Change between baseline and 9 months after entry
  weighted frequency of intentional communication from the Communication and Symbolic Behavior Scale, high is good range is 0 - 400

SECONDARY OUTCOMES:
Growth in play | Change from Baseline to 9 months after entry
  raw scores from Developmental Play Assessment, high is good, range is 0 to 50
Motor imitation | Change from Baseline to 9 months after entry
  raw scores from the Structured Social Imitation Scale, high is good, range 0 - 50
Autism social affect symptomatology | 9 months after entry
  average of z score from raw scores from Communication and Symbolic Behavior Scale and Autism Diagnositic Observation Schedule (reflected) if they are correlated > .4, after reflection high is good, -4 to 4
Language delay | 9 months after entry
  average of z scores from standard scores or percentile rankings from MacAuthur Communication Development Index and Mullen Scale of Early Learning if they are correlated above .4, high is good, range is -4 to 4
language level | Change from baseline to 9 mos after treatment ends
  average of time 4-referenced z scores from raw scores from Communication and Symbolic Behavior Scales, Brief Observation of Social Communication Change, and MacArthur Communication Development Index if they are correlated above .4, High is good, -4 to 4
parent implementation of ImPACT treatment | change from baseline to immediately post-treatment
  fidelity of treatment of aspects of ImPACT treatment from PCS and PCFP

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Yoder, Ph.D., Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Vanderbilt University, Nashville, Tennessee
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No